CLINICAL TRIAL: NCT00446550
Title: A Randomized, Open-label Study To Assess the Safety and Tolerability of AT2101 in Treatment-naive Adult Patients With Type 1 Gaucher Disease
Brief Title: A Study of Oral AT2101 (Afegostat Tartrate) in Treatment-naive Patients With Gaucher Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAU-CL-202
Record Dates: First submitted 2007-03-09; First posted 2007-03-13 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Gaucher Disease; Type 1 Gaucher Disease; Gaucher Disease, Type 1
Keywords: Amicus Therapeutics; afegostat tartrate; isofagomine tartrate; AT2101
MeSH Terms: conditions — Gaucher Disease | interventions — AT2101

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Afegostat Tartrate Treatment Regimen 1 (Experimental): For the first 2 weeks, afegostat tartrate was administered orally at a dose of 225 milligrams (mg) once daily (QD) for 7 consecutive days, followed by no study medication for 7 consecutive days. After 2 weeks, participants then took 225 mg afegostat tartrate QD for 3 consecutive days, followed by no study medication for 4 consecutive days. This 3-days-on/4-days-off treatment regimen was followed for 22 weeks.
  Interventions: Drug: afegostat tartrate
- Afegostat Tartrate Treatment Regimen 2 (Experimental): Afegostat tartrate was administered orally at a dose of 225 mg QD for 7 consecutive days, followed by no study medication for 7 consecutive days. This 7-days-on/7-days-off treatment regimen was followed for 24 weeks.
  Interventions: Drug: afegostat tartrate

INTERVENTIONS:
Drug: afegostat tartrate
  Other Names: isofagomine tartrate; AT2101

SUMMARY:
This study evaluated the safety and tolerability of afegostat tartrate in participants with type 1 Gaucher disease who were not receiving enzyme replacement therapy (ERT) or substrate reduction therapy (SRT).

DETAILED DESCRIPTION:
This was a Phase 2, open-label study in participants with Gaucher disease, a lysosomal storage disorder. Afegostat tartrate (also known as AT2101 or isofagomine tartrate) is designed to act as a pharmacological chaperone by selectively binding to misfolded β-glucocerebrosidase (GCase) and helping it fold correctly, intended to restore GCase activity. The study consisted of a 21-day screening period, a 24-week treatment period, and follow-up visit (Day 183, end-of-study). Participants were randomized in a 1:1 ratio to 1 of 2 treatment regimens for afegostat tartrate (3 days on treatment/4 days off or 7 days on treatment/7 days off).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of type 1 Gaucher disease with a known genotype and a documented missense gene mutation in at least 1 of the 2 gene-encoding β-glucosidase (GBA) alleles
* Clinically stable
* Treatment naïve to ERT and SRT or had not received ERT or SRT in the 12 months before screening
* Willing to not initiate ERT or SRT treatment during study participation
* Male or female participants, 18 to 74 years old, inclusive
* At the screening period (Day -21 to Day -1), participants must have met at least 2 of the following criteria: platelet count of ≤150,000 per microliter, hemoglobin ≤12 grams/deciliter (g/dL) for females and ≤13 g/dL for males, liver volume ≥1.25 multiples of normal (MN), and spleen volume ≥2 MN
* All participants of reproductive potential were required to practice an acceptable method of contraception
* Provided written informed consent to participate in the study

Exclusion Criteria:

* A clinically significant disease other than Gaucher disease, severe complications from Gaucher disease, or serious intercurrent illness that precluded participation in the study in the opinion of the investigator
* During the screening period, had any clinically significant findings as deemed by the investigator
* Partial or total splenectomy
* Documentation of moderate or severe pulmonary hypertension, defined as pulmonary arterial pressure >35 millimeters of mercury (mmHg) or significant Gaucher-related lung disease
* History of allergy or sensitivity to the study drug or any excipients, including any prior serious allergic reaction to iminosugars
* Pacemaker or other contraindication for magnetic resonance imaging (MRI) scanning
* Pregnant or breast-feeding
* Current/recent drug or alcohol abuse
* Treatment with any investigational product in the last 90 days before study entry
* Treatment in the previous 90 days with any drug known to have a well-defined potential for toxicity to a major organ
* Presence of symptoms of gastrointestinal, liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-06-11 (Actual); Primary Completion 2009-08-20 (Actual); Study Completion 2009-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — Amicus Therapeutics
Locations (11):
- United States (7):
  - Beverly Hills, California
  - Coral Springs, Florida
  - Decatur, Georgia
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Boston, Massachusetts
  - Cincinnati, Ohio
- Israel (2):
  - Haifa
  - Tel Aviv
- Johannesburg, South Africa
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Confirmatory β-glucosidase (GBA) genotype testing was done at screening to confirm reported genotype (with the exception of participants enrolled in Israel).19 participants received at least 1 dose of study drug. All participants were eligible for inclusion in both the safety and the pharmacodynamics (PD) populations.
Period: Overall Study
Arm/Group | Afegostat Tartrate Treatment Regimen 1 | Afegostat Tartrate Treatment Regimen 2
Started | 11 | 8
Safety Population (All participants who received at least 1 dose of study drug.) | 11 | 8
PD Population (Participants in the Safety Population with a baseline and at least 1 post-baseline PD measurement.) | 11 | 8
Completed | 10 | 8
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Afegostat Tartrate Treatment Regimen 1: For the first 2 weeks, afegostat tartrate was administered orally at a dose of 225 mg QD for 7 consecutive days, followed by no study medication for 7 consecutive days. After 2 weeks, participants then took 225 mg afegostat tartrate QD for 3 consecutive days, followed by no study medication for 4 consecutive days. This 3-days-on/4-days-off treatment regimen was followed for 22 weeks.
- Total: Total of all reporting groups
Arm/Group | Afegostat Tartrate Treatment Regimen 1 | Afegostat Tartrate Treatment Regimen 2 | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (16.27) | 39.1 (17.62) | 41.4 (16.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Who Experienced Severe Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any adverse event (AE) with start date on or after administration of study drug or pre-existing conditions that worsened on or after the start of the first study drug administration (on Day 1). A severe AE defined as an AE that was incapacitating and required medical intervention. The number of participants who experienced 1 or more severe TEAEs after dosing on Day 1 through the end of follow-up (Day 183) is presented. A summary of serious and all other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 (after dosing) through Day 183
Population: Safety Population: all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Afegostat Tartrate Treatment Regimen 2: Afegostat tartrate was administered orally at a dose of 225 mg QD for 7 consecutive days followed by no study medication for 7 consecutive days. This 7-days-on/7-days-off treatment regimen was followed for 24 weeks.
Arm/Group | Afegostat Tartrate Treatment Regimen 1 | Afegostat Tartrate Treatment Regimen 2
Number analyzed (Participants) | 11 | 8
Participants | 2 | 0

2. Secondary Outcome: Change From Baseline To End Of Treatment In β-glucocerebrosidase (GCase) Levels In White Blood Cells (WBC)
Description: GCase is a biomarker used to assess the PD effects of afegostat tartrate. Blood samples were collected to assess GCase levels in WBC. The baseline value was defined as the last non-missing value before the start of study drug.
Time Frame: Baseline, Day 169
Population: PD Population: all participants who were included in the Safety Population and had a baseline and at least 1 post-baseline PD measurement.
Measure: Mean (Standard Deviation); unit: picomole/minute/mg
Arm/Group | Afegostat Tartrate Treatment Regimen 1 | Afegostat Tartrate Treatment Regimen 2
Number analyzed (Participants) | 11 | 7
picomole/minute/mg | 10.2 (15.87) | 3.9 (4.12)

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) to Day 183
Arm/Group | Afegostat Tartrate Treatment Regimen 1 | Afegostat Tartrate Treatment Regimen 2
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/8
Other Adverse Events (participants affected / at risk) | 10/11 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Afegostat Tartrate Treatment Regimen 1 (N=11) | Afegostat Tartrate Treatment Regimen 2 (N=8)
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Abnormal sensation in eye (Eye disorders) | 1 | 1
Chalazion (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Conjunctival irritation (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 2
Eye inflammation (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 2 | 1
Eye pruritus (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 3 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Adverse drug reaction (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Eyelid infection (Infections and infestations) | 0 | 1
Fungal rash (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Bacteria urine (Investigations) | 0 | 1
Vitamin B12 decreased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Poor quality sleep (Nervous system disorders) | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 1/4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can publish only the results from this trial, provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review prior to submission for publication. If requested and prior to publication, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication for an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.